CLINICAL TRIAL: NCT05745142
Title: A Retrospective Registry Based Study for Evaluating Treatment Response in Patients Targeted Treated With Metastatic Renal Cell Carcinoma (mRCC) With Sunitinib in First-line Therapy
Brief Title: A Study to go Back Into Records and Observe How People With Metastatic Renal Cell Carcinoma (mRCC) Who Received a Medicine Called Sunitinib Responded to This Medicine.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181235
Record Dates: First submitted 2023-01-26; First posted 2023-02-27 (Actual); Results first posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-02

CONDITIONS: Carcinoma, Renal Cell; Clear-cell Metastatic Renal Cell Carcinoma
Keywords: mRCC; Metastatic Renal Cell Carcinoma; Clear-cell metastatic renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Clear-cell metastatic renal cell carcinoma | interventions — Sunitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- metastatic Renal Cell Carcinoma patients: metastatic Renal Cell Carcinoma patients with clear cell histology.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — as provided in real world practice

SUMMARY:
The purpose of this study is to understand how patients with mRCC respond to the study medicine (called sunitinib) when they receive it as the first line of treatment after finding out the cause for the disease.

This study will look into how different and how well groups of people with high chances of developing the disease respond to the study medicine.

All data for this study will be anonymously extracted from data already entered in RCC Registry which is owned by Turkish Oncology Group Association (TOGD).

This study will pull out records from the Registry between 01-Mar-2019 and 30-Oct-2022 that belongs to people:

* who are Turkish citizens
* who are older than 18 years
* who were found out to have mRCC
* who received sunitinib as the first line treatment after finding out the cause for the disease

This study will look at the responses, experiences and how long the patients use the study medicine sunitinib.

DETAILED DESCRIPTION:
This study is designed as a local, non-interventional, retrospective, registry-based study to observe treatment response in patients with metastatic Renal Cell Carcinoma with Sunitinib First-Line Therapy based on data extracted and analyzed from the RCC Registry.

The annual disease burden in contributing centers to RCC Registry is approximately 100 patient/center, the treatment of an average of 250 patients per year is continued in the centers. Therefore, it is estimated that information of approximately 400 eligible patients who were registered in RCC Registry from 2019 to 2022 will be included in the analysis.

RCC Registry will be used as the sole data source for this study. For this purpose, no Case Report Forms (CRFs) or Data Collection Tools (DCTs) will be utilized, but the RCC Registry database will be used directly. Eligible patients' data will be anonymized and extracted for analysis by the registry owner, for this study.

ELIGIBILITY:
Inclusion Criteria:

* Being a Turkish citizen.
* Being older than 18 years-old.
* Being clinically diagnosed with mRCC and treated.
* Being treated with Sunitinib in first line

Exclusion Criteria:

* Patients whose treatment was initiated but excluded from follow-up for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RCC Registry will be screened for all patients who meets all inclusion criteria and who doesn't meet the exclusion criterion defined in the study protocol and who were treated with Sunitinib in first-line therapy for mRCC and were registered to the database between 2019 and 2022.
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A6181235

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with metastatic renal cell carcinoma (mRCC), who were being treated with Sunitinib in first-line therapy and got registered in RCC database between 01-March-2019 and 30-October-2022 were included in this study and their data was observed retrospectively.
Pre-assignment Details: RCC registry was a data log where clinical information was recorded by inviting participants who met the selection criteria according to protocol (Turkish citizen, older than 18 years, being diagnosed with mRCC and being treated with sunitinib in first line). It was used as data source for this study and the participant data was retrospectively recorded in the study database. A total of 376 participants were included in this study which pulled out records from the RCC registry.
Groups:
- Sunitinib: Participants diagnosed with mRCC, who were being treated with Sunitinib as first-line therapy in real world practice and who got registered in RCC registry in Turkey were included. The recommended dose of sunitinib in mRCC is 50 milligrams (mg) orally daily for 4 weeks, followed by 2 weeks off treatment (4/2 schedule).
Period: Overall Study
Arm/Group | Sunitinib
Started | 376
Completed | 376
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Groups:
- Sunitinib: Participants diagnosed with mRCC on treatment with Sunitinib as first-line therapy in real world practice and were registered in RCC registry in Turkey were included. The recommended dose of sunitinib in mRCC is 50 mg orally daily for 4 weeks, followed by 2 weeks off treatment (4/2 schedule).
Arm/Group | Sunitinib
Number analyzed (Participants) | 376
Age, Continuous [Median (Full Range); unit: Years] | 58 [53 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95
  Male | 281
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of Participants With Comorbidities [Count of Participants; unit: Participants]
  Hypertension | 154
  Diabetes Mellitus | 81
Number of Participants According to Previous Nephrectomy Status [Count of Participants; unit: Participants]
  Yes | 288
  No | 83
  Missing | 5
Number of Participants According to Previous Interferon Use [Count of Participants; unit: Participants]
  Yes | 189
  No | 187
Number of Participants According to International Metastatic RCC Database Consortium (IMDC) Groups [Count of Participants; unit: Participants] — IMDC criteria had 6 risk factors: Karnofsky Performance Status (KPS) less than (<) 80% (ability to perform ordinary tasks, 0 [dead] -100 [normal]); time from diagnosis to start of systemic therapy <1 year; corrected serum calcium; neutrophils and platelets more than (>) upper limit of normal (ULN); hemoglobin <lower limit of normal (LLN). Present risk factors were added, and then participants were stratified as: favorable (0 factor), intermediate (1-2 factors), poor (more than or equal to [>=]3 factors).
  Participants
    Favorable | 70
    Intermediate | 168
    Poor | 73
    Missing | 65
Number of Participants According to Memorial Sloan-Kettering Cancer Center (MSKCC) Groups [Count of Participants; unit: Participants] — MSKCC criteria had 5 risk factors: KPS <80% (ability to perform ordinary tasks, 0 [dead] -100 [normal]); time from diagnosis to start of systemic therapy <12 months; hemoglobin <LLN; lactate dehydrogenase 1.5*ULN; corrected serum calcium >10 milligram per deciliter (mg/dL). Present risk factors were added, and participants were stratified as: favorable (0 factor), intermediate (1-2 factors), poor (>=3 factors).
  Participants
    Favorable | 62
    Intermediate | 162
    Poor | 37
    Missing | 115
Number of Participants According to Metastatic Sites [Count of Participants; unit: Participants] — Participants could have more than 1 metastatic sites.
  Participants
    Lung | 295
    Bone | 172
    Liver | 80
    Central Nervous System | 50
Number of Participants According to Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Grade 0: fully active, able to carry on all pre-disease performance without restriction; Grade 1: restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, Grade 2: ambulatory and capable of all self-care, but unable to carry out any work activities, up and about more than 50% of waking hours, Grade 3: capable of only limited self-care, confined to bed or chair for more than 50% of waking hours, Grade 4: completely disabled; cannot carry on any self-care; totally confined to bed or chair.
  Participants
    0-1 | 271
    2 | 69
    3-4 | 12
    Missing | 24
Number of Participants According to Initial Tumor, Node, Metastasis (TNM) Stage [Count of Participants; unit: Participants] — 0= tumor is 7 centimeter (cm) across, is only in kidney and has not spread; 1= tumor is larger than 7 cm across, is only in kidney and has not spread; 2= tumor grown into a major vein, not growing into adrenal gland or beyond Gerota's fascia and has not spread; 3= tumor is of any size, not spread beyond Gerota's fascia and has not spread; 4= tumor is growing beyond Gerota's fascia and may/may not has spread. The higher the number, the larger the tumor and/or the more it has spread into nearby tissues.
  Participants
    1 | 32
    2 | 43
    3 | 52
    4 | 191
    Missing | 58

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) According to Disease Risk Group in IMDC
Description: ORR: percentage of participants with partial response (PR) and complete response (CR). As per response evaluation criteria in solid tumors (RECIST)1.1 criteria: CR = disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis); PR = at least 30% decrease in sum of diameters of target lesions taking as reference baseline sum diameters. IMDC assessed as favorable (0), intermediate (1-2) or poor (>=3) based on number of criteria present (KPS <80%; time from diagnosis to start of systemic therapy <1 year; corrected serum calcium [Ca]; neutrophils and platelets >ULN; hemoglobin [hg] <LLN).
Time Frame: From initiation of sunitinib treatment (retrospective data) till PR and CR or death or progression (up to 30-Oct-2022, cut-off for data registry); approximate follow-up duration of 73 months [from data extracted from registry database]
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study. Here, "Number of Participants Analyzed" signified participants who were evaluable for this outcome measure and with non-missing data; "Number Analyzed" signified participants evaluable for specified rows.
Measure: Number; unit: Percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 132
Percentage of participants
  Favorable: number analyzed (Participants) | 33
  Favorable | 57.5
  Intermediate: number analyzed (Participants) | 74
  Intermediate | 44.6
  Poor: number analyzed (Participants) | 25
  Poor | 24.0

2. Primary Outcome: Response Rates According to Disease Risk Group in IMDC
Description: RECIST1.1- CR: disappearance of all lesions & normalization of tumor marker level. Any pathological lymph nodes must have reduction in short axis to <10 mm. All lymph nodes must be non-pathological in size (<10 mm short axis); PR: at least 30% decrease in sum of diameters of target lesions taking as reference baseline sum diameters; progressive disease (PD): at least 20% increase in sum of longest dimensions of target lesions, reference to the smallest sum of the longest dimensions recorded since treatment started, or appearance of 1 or more new lesions or increase of at least 5 mm in addition to the relative increase of 20%; stable disease (SD): neither shrinkage for CR/PR nor increase for PD taking as reference smallest sum of longest diameters since treatment start. IMDC: favorable (0), intermediate (1-2) or poor (>=3) based on number of criteria present (KPS <80%; time from diagnosis to start of systemic therapy <1 year; corrected serum Ca]; neutrophils & platelets >ULN; hg <LLN).
Time Frame: From initiation of sunitinib treatment (retrospective data) till PR/ CR/ SD/ death or progression (up to 30-Oct-2022, cut-off for data registry); approximate follow-up duration of 73 months [from data extracted from registry database]
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 132
Percentage of participants
  CR: Favorable: number analyzed (Participants) | 33
  CR: Favorable | 3.0
  CR: Intermediate: number analyzed (Participants) | 74
  CR: Intermediate | 5.4
  CR: Poor: number analyzed (Participants) | 25
  CR: Poor | 4.0
  PR: Favorable: number analyzed (Participants) | 33
  PR: Favorable | 54.5
  PR: Intermediate: number analyzed (Participants) | 74
  PR: Intermediate | 39.2
  PR: Poor: number analyzed (Participants) | 25
  PR: Poor | 20.0
  SD: Favorable: number analyzed (Participants) | 33
  SD: Favorable | 18.2
  SD: Intermediate: number analyzed (Participants) | 74
  SD: Intermediate | 32.4
  SD: Poor: number analyzed (Participants) | 25
  SD: Poor | 36.0
  PD: Favorable: number analyzed (Participants) | 33
  PD: Favorable | 24.2
  PD: Intermediate: number analyzed (Participants) | 74
  PD: Intermediate | 23.0
  PD: Poor: number analyzed (Participants) | 25
  PD: Poor | 40.0

3. Primary Outcome: ORR According to Disease Risk Group in MSKCC
Description: ORR: percentage of participants with PR and CR. As per RECIST 1.1 criteria: CR = disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis); PR = at least 30% decrease in sum of diameters of target lesions taking as reference baseline sum diameters. MSKCC assessed as favorable (0), intermediate (1-2) or poor (>=3) based on number of criteria present [KPS <80%, time from diagnosis to start of systemic therapy <12 months, lactate dehydrogenase >1.5*ULN, hemoglobin <LLN, serum calcium >10 mg/dL].
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 108
Percentage of participants
  Favorable: number analyzed (Participants) | 30
  Favorable | 66.6
  Intermediate: number analyzed (Participants) | 68
  Intermediate | 44.1
  Poor: number analyzed (Participants) | 10
  Poor | 30

4. Primary Outcome: Response Rates According to Disease Risk Group in MSKCC
Description: RECIST1.1- CR: disappearance of all lesions and normalization of tumor marker level. Any pathological lymph nodes must have reduction in short axis to <10 mm. All lymph nodes must be non-pathological in size (<10 mm short axis); PR: at least 30% decrease in sum of diameters of target lesions taking as reference baseline sum diameters; PD: at least 20% increase in sum of longest dimensions of target lesions, reference to the smallest sum of the longest dimensions recorded since treatment started, or the appearance of 1 or more new lesions or increase of at least 5 mm in addition to the relative increase of 20%; SD: neither shrinkage for CR/PR nor increase for PD taking as reference smallest sum of longest diameters since treatment start. MSKCC assessed as favourable (0), intermediate (1-2) or poor (>=3) based on number of criteria present [KPS <80%, time from diagnosis to start of systemic therapy <12 months, lactate dehydrogenase >1.5*ULN, hemoglobin <LLN, serum calcium >10 mg/dL].
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 108
Percentage of participants
  CR: Favorable: number analyzed (Participants) | 30
  CR: Favorable | 3.3
  CR: Intermediate: number analyzed (Participants) | 68
  CR: Intermediate | 2.9
  CR: Poor: number analyzed (Participants) | 10
  CR: Poor | 0.0
  PR: Favorable: number analyzed (Participants) | 30
  PR: Favorable | 63.3
  PR: Intermediate: number analyzed (Participants) | 68
  PR: Intermediate | 41.2
  PR: Poor: number analyzed (Participants) | 10
  PR: Poor | 30.0
  SD: Favorable: number analyzed (Participants) | 30
  SD: Favorable | 16.7
  SD: Intermediate: number analyzed (Participants) | 68
  SD: Intermediate | 25.0
  SD: Poor: number analyzed (Participants) | 10
  SD: Poor | 30.0
  PD: Favorable: number analyzed (Participants) | 30
  PD: Favorable | 16.7
  PD: Intermediate: number analyzed (Participants) | 68
  PD: Intermediate | 30.9
  PD: Poor: number analyzed (Participants) | 10
  PD: Poor | 40.0

5. Secondary Outcome: Overall Survival (OS) Rate According to Disease Risk Group in IMDC
Description: OS was defined as the time from the start of the treatment until the date of death. If no death was recorded, data was censored at latest available date in data. IMDC assessed as favorable (0), intermediate (1-2) or poor (>=3) based on number of criteria present (KPS <80%; time from diagnosis to start of systemic therapy <1 year; corrected serum Ca; neutrophils and platelets >ULN; hg <LLN).
Time Frame: From initiation of sunitinib treatment (retrospective data) till death or censored date (up to 30-Oct-2022, cut-off for data registry); approximate follow-up duration of 73 months [from data extracted from registry database]
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study. Here, "Number of Participants Analyzed" signified participants with non-missing data and "Number Analyzed" signified participants evaluable for specified rows.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib
Number analyzed (Participants) | 311
Months
  Favorable: number analyzed (Participants) | 70
  Favorable | 41.9 [24.9 to 58.9]
  Intermediate: number analyzed (Participants) | 168
  Intermediate | 31.2 [21.8 to 40.6]
  Poor: number analyzed (Participants) | 73
  Poor | 7.1 [3.9 to 10.3]

6. Secondary Outcome: Progression-Free Survival (PFS) According to Disease Risk Group in IMDC
Description: PFS: duration from start of treatment to disease progression (PD), end of treatment date or date of death. PD: at least 20% increase in sum of longest dimensions of target lesions, reference to the smallest sum of the longest dimensions recorded since treatment started, or the appearance of 1 or more new lesions or increase of at least 5 mm in addition to the relative increase of 20%. IMDC assessed as favorable (0), intermediate (1-2) or poor (>=3) based on number of criteria present (KPS <80%; time from diagnosis to start of systemic therapy <1 year; corrected serum Ca; neutrophils and platelets >ULN; hg <LLN).
Time Frame: From initiation of sunitinib treatment (retrospective data) till progression end of treatment date or date of death (up to 30-Oct-2022, cut-off for data registry); approximate follow-up duration of 73 months [from data extracted from registry database]
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib
Number analyzed (Participants) | 311
Months
  Favorable: number analyzed (Participants) | 70
  Favorable | 19.4 [11.6 to 27.4]
  Intermediate: number analyzed (Participants) | 168
  Intermediate | 13.14 [10.0 to 16.2]
  Poor: number analyzed (Participants) | 73
  Poor | 5.02 [4.1 to 5.9]

7. Secondary Outcome: OS According to Disease Risk Group in MSKCC
Description: OS was defined as the time from the start of the treatment until the date of death. If no death was recorded, data was censored at latest available date in data. MSKCC assessed as favourable (0), intermediate (1-2) or poor (>=3) based on number of criteria present [KPS <80%, time from diagnosis to start of systemic therapy <12 months, lactate dehydrogenase >1.5*ULN, hemoglobin <LLN, serum calcium >10 mg/dL].
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib
Number analyzed (Participants) | 261
Months
  Favorable: number analyzed (Participants) | 62
  Favorable | 52.2 [31.8 to 72.7]
  Intermediate: number analyzed (Participants) | 162
  Intermediate | 24.0 [13.9 to 34.1]
  Poor: number analyzed (Participants) | 37
  Poor | 4.9 [3.6 to 6.8]

8. Secondary Outcome: PFS According to Disease Risk Group in MSKCC
Description: PFS: duration from start of treatment to PD, end of treatment date or date of death. PD: at least 20% increase in sum of longest dimensions of target lesions, reference to the smallest sum of the longest dimensions recorded since treatment started, or the appearance of 1 or more new lesions or increase of at least 5 mm in addition to the relative increase of 20%. MSKCC assessed as favourable (0), intermediate (1-2) or poor (>=3) based on number of criteria present [KPS <80%, time from diagnosis to start of systemic therapy <12 months, lactate dehydrogenase >1.5*ULN, hemoglobin <LLN, serum calcium >10 mg/dL].
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib
Number analyzed (Participants) | 261
Months
  Favorable: number analyzed (Participants) | 62
  Favorable | NA [NA to NA] — In RCC registry, data was not available for PFS per MSKCC risk categories, hence could not be reported.
  Intermediate: number analyzed (Participants) | 162
  Intermediate | NA [NA to NA] — In RCC registry, data was not available for PFS per MSKCC risk categories, hence could not be reported.
  Poor: number analyzed (Participants) | 37
  Poor | NA [NA to NA] — In RCC registry, data was not available for PFS per MSKCC risk categories, hence could not be reported.

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not planned to be collected during the study.
Description: Minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) could not be met. Hence, adverse events were not collected and reported.
Arm/Group | Sunitinib
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/42/NCT05745142/Prot_SAP_000.pdf